CLINICAL TRIAL: NCT02197728
Title: Comparing Two Devices of Uterine Manipulation and Vaginal Fornix Delineation at Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-326
Record Dates: First submitted 2014-05-23; First posted 2014-07-23 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Laparoscopic Hysterectomy for Benign Conditions
Keywords: hysterectomy, uterine manipulator, thermal damage, laparoscopy, colpotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hohl uterine manipulator ® (Active Comparator): Total laparoscopic hysterectomy is performed using the Hohl uterine manipulator ®
  Interventions: Device: Use of the Colpo-Probe™ Vaginal Fornix Delineator or Hohl manipulator® during total laparoscopic hysterectomy
- Colpo-Probe™ Vaginal Fornix Delineator (Active Comparator): Total laparoscopic hysterectomy is performed using the Colpo-Probe™ Vaginal Fornix Delineator
  Interventions: Device: Use of the Colpo-Probe™ Vaginal Fornix Delineator or Hohl manipulator® during total laparoscopic hysterectomy

INTERVENTIONS:
Device: Use of the Colpo-Probe™ Vaginal Fornix Delineator or Hohl manipulator® during total laparoscopic hysterectomy

SUMMARY:
We hypothesize, that the use of the Hohl manipulator® at total laparoscopic hysterectomy reduces operative time (from skin incision to detachment of the uterus) and lateral termal damage of the vaginal wall during colpotomy due to the following reasons: (1) Uterine manipulation is better with the Hohl manipulator®, thereby facilitating dissection during all aspects of the surgery, (2) more tension can be applied on the vagina during colpotomy, thereby hastening electrosurgical transection, reducing activation time and reduce lateral thermal damage and (3) tension on the vagina can be applied until the colpotomy is finished, due to the tight connection between the Hohl manipulator® and the cervix of the uterus, which also affects speed of transection, electrosurgical device activation time and lateral thermal damage.

ELIGIBILITY:
Inclusion Criteria:

* All women aged over 18 years, scheduled for a laparoscopic hysterectomy for a benign disorder will be asked to participate and included after written informed consent.

Exclusion Criteria:

* pregnancy
* malignancy
* if uterine size exceeds 20 weeks of gestation
* or if the uterus could be removed by a vaginal approach

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Detachment of the uterus | 45 minutes to 3 hours
  Operative time from skin incision to detachment of uterus. Times are routinely collected by operating room nursing staff.
Thermal Damage | 2 weeks post surgery
  Lateral thermal damage to the vagina will be measured on the specimen (in mm) at the time of pathologic evaluation.
Colpotomy | 3 minutes to 20 minutes
  Time from first monopolar energy activation to completion of colpotomy. Operative times are routinely collected by operating room nursing staff.

SECONDARY OUTCOMES:
Blood Loss | 45 minutes to 3 hours
  Total amount of blood lost throughout surgery. Measured in cc.
Pain | 24h post surgery
  Amount of post operative pain measured using a pain sensitivity scale.
Manipulator Installment | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Guylaine Lefebvre, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael´s Hospital, Toronto, Ontario, Canada